CLINICAL TRIAL: NCT03489967
Title: Treatment of Mild-to-moderate Hypoglycemia in Adults With Type 1 Diabetes: a Validation Study
Brief Title: Treatment of Hypoglycemia in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HYPO-T
Record Dates: First submitted 2018-03-09; First posted 2018-04-06 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Type 1 Diabetes
Keywords: Hypoglycemia, carbohydrates
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 16g of carbohydrates - Glucose levels < 3.0 mmol/L (Active Comparator): Hypoglycemia treatment with 16g of carbohydrates will be given when glucose levels are below 3.0 mmol/L.
  Interventions: Other: Induced-hypoglycemia test
- 16g of carbohydrates - Glucose levels 3.0-3.5 mmol/L (Active Comparator): Hypoglycemia treatment with 16g of carbohydrates will be given when glucose levels are between 3.0 and 3.5 mmol/L.
  Interventions: Other: Induced-hypoglycemia test
- 32g of carbohydrates - Glucose levels < 3.0 mmol/L (Active Comparator): Hypoglycemia treatment with 32g of carbohydrates will be given when glucose levels are below 3.0 mmol/L
  Interventions: Other: Induced-hypoglycemia test
- 32g of carbohydrates - Glucose levels 3.0-3.5 mmol/L (Active Comparator): Hypoglycemia treatment with 32g of carbohydrates will be given when glucose levels are between 3.0 and 3.5 mmol/L.
  Interventions: Other: Induced-hypoglycemia test

INTERVENTIONS:
Other: Induced-hypoglycemia test — Participants will be admitted at the research center at 7:00 after an overnight fast. A venous catheter will be inserted into an arm vein for blood sampling purposes. A subcutaneous insulin bolus will be administered to induce hypoglycemia. Oral treatment (16g of carbohydrates or 32g of carbohydrates) will be given when plasma glucose levels are at the target threshold of < 3.0 mmol/L or 3.0-3.5 mmol/L. Hypoglycemia symptoms will be assessed every 10 minutes by the participant using a validated scale starting from the time of insulin bolus until hypoglycemia recovery. One hour after hypoglycemia recovery, a standardized meal will be given.

SUMMARY:
According to guidelines, when a mild-to-moderate hypoglycemia occurs (capillary blood glucose < 4.0 mmol/L), 15-20g of rapidly absorbed carbohydrates should be ingested. Patients should re-test and re-ingest 15-20g carbohydrates every 15 minutes until they recover from hypoglycemia. These recommendations were principally based on two studies conducted in the 80s before the introduction of intensive insulin therapy secondary to the DCCT trial and with insulin formulations with largely different pharmacokinetic profiles from current insulin analogs. Recent studies suggest that with current insulin analogs and intensive therapeutic approach, 15g of carbohydrates may be insufficient to rapidly correct an important proportion of hypoglycemic episodes. It is thus important to determine if the recommended hypoglycemia treatment remains the recommendation.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. Treatment with multiple daily insulin injections or insulin pump therapy and using insulin analogs (rapid, ultra-rapid and basal).
4. HbA1c ≤ 10%.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Known significant cardiac rhythm abnormality based on investigator judgment.
4. Abnormal blood panel and/or anemia (Hb < 100g/L).
5. Ongoing pregnancy or breastfeeding.
6. Severe hypoglycemic episode within 1 month of screening.
7. Known uncorrected hypokalemia (potassium < 3.5 mmol/L; available within the past 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in glucose levels 15 minutes after hypoglycemic treatment | 15 minutes after hypoglycemic treatment
  Change in glucose levels 15 minutes after hypoglycemic treatment (16g vs. 32g of carbohydrates) when glucose levels at the time of treatment are below 3.0 mmol/L or between 3.0 and 3.5 mmol/L.

SECONDARY OUTCOMES:
Change in glucose levels 20 minutes after hypoglycemic treatment | 20 minutes after hypoglycemic treatment
  Change in glucose levels 20 minutes after hypoglycemic treatment (16g vs. 32g of carbohydrates) when glucose levels at the time of treatment are below 3.0 mmol/L or between 3.0 and 3.5 mmol/L.
Change in glucose levels 30 minutes after hypoglycemic treatment | 30 minutes after hypoglycemic treatment
  Change in glucose levels 30 minutes after hypoglycemic treatment (16g vs. 32g of carbohydrates) when glucose levels at the time of treatment are below 3.0 mmol/L or between 3.0 and 3.5 mmol/L.
Change in glucose levels 45 minutes after hypoglycemic treatment | 45 minutes after hypoglycemic treatment
  Change in glucose levels 45 minutes after hypoglycemic treatment (16g vs. 32g of carbohydrates) when glucose levels at the time of treatment are below 3.0 mmol/L or between 3.0 and 3.5 mmol/L.
Change in glucose levels 60 minutes after hypoglycemic treatment | 60 minutes after hypoglycemic treatment
  Change in glucose levels 60 minutes after hypoglycemic treatment (16g vs. 32g of carbohydrates) when glucose levels at the time of treatment are below 3.0 mmol/L or between 3.0 and 3.5 mmol/L.
Number of participants with glucose levels above 8.0 mmol/L 1 hour after hypoglycemia correction | 60 minutes after hypoglycemia correction
Number of participants with glucose levels above 10.0 mmol/L 1 hour after hypoglycemia correction | 60 minutes after hypoglycemia correction
Glucose levels 60 minutes after meal consumption | 60 minutes after meal consumption
Glucose levels 90 minutes after meal consumption | 90 minutes after meal consumption
Number of patients for whom hypoglycemia was corrected 10 minutes after hypoglycemic treatment | 10 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia was corrected 15 minutes after hypoglycemic treatment | 15 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia was corrected 20 minutes after hypoglycemic treatment | 20 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia was corrected 25 minutes after hypoglycemic treatment | 25 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia was corrected 30 minutes after hypoglycemic treatment | 30 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia was corrected 35 minutes after hypoglycemic treatment | 35 minutes after hypoglycemic treatment
Number of hypoglycemic events corrected 10 minutes after hypoglycemic treatment | 10 minutes after hypoglycemic treatment
Number of hypoglycemic events corrected 15 minutes after hypoglycemic treatment | 15 minutes after hypoglycemic treatment
Number of hypoglycemic events corrected 20 minutes after hypoglycemic treatment | 20 minutes after hypoglycemic treatment
Number of hypoglycemic events corrected 25 minutes after hypoglycemic treatment | 25 minutes after hypoglycemic treatment
Number of hypoglycemic events corrected 30 minutes after hypoglycemic treatment | 30 minutes after hypoglycemic treatment
Number of hypoglycemic events corrected 35 minutes after hypoglycemic treatment | 35 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia symptoms disappeared 10 minutes after hypoglycemic treatment | 10 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia symptoms disappeared 15 minutes after hypoglycemic treatment | 15 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia symptoms disappeared 20 minutes after hypoglycemic treatment | 20 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia symptoms disappeared 25 minutes after hypoglycemic treatment | 25 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia symptoms disappeared 30 minutes after hypoglycemic treatment | 30 minutes after hypoglycemic treatment
Number of patients for whom hypoglycemia symptoms disappeared 35 minutes after hypoglycemic treatment | 35 minutes after hypoglycemic treatment
Number of patients requiring a second treatment 40 minutes after the first hypoglycemic treatment | 40 minutes after the first hypoglycemic treatment
Number of patients requiring a second treatment 15 minutes after the first hypoglycemic treatment | 15 minutes after the first hypoglycemic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Canada

REFERENCES:
- [Derived] Taleb N, Gingras V, Cheng R, Parent V, Messier V, Bovan D, Shohoudi A, Brazeau AS, Rabasa-Lhoret R. Non-severe hypoglycemia in type 1 diabetes: a randomized crossover trial comparing two quantities of oral carbohydrates at different insulin-induced hypoglycemia ranges. Front Endocrinol (Lausanne). 2023 Jun 2;14:1186680. doi: 10.3389/fendo.2023.1186680. eCollection 2023. PMID 37334295